CLINICAL TRIAL: NCT03185208
Title: Evaluation of Brain and Cognitive Changes in Older Adults With MCI Taking Lithium to Prevent Alzheimer Type Dementia
Brief Title: Lithium As a Treatment to Prevent Impairment of Cognition in Elders
Acronym: LATTICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ariel Gildengers, MD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Ariel Gildengers, MD, Associate Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO17030527; R01AG055389-01 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-06-14 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Lithium; Mild Cognitive Impairment; MCI; Dementia; Alzheimer; Alzheimer's Disease; Cognition; Memory; Thinking; Prevention; amyloid; imaging; MRI; PET; tau; plaques; tangles
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Pick Disease of the Brain; Plaque, Amyloid | interventions — Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: Longitudinal, randomized, double-blind, placebo-controlled experimental trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators (who will also be prescribers/care providers), and both clinical and cognitive raters will be blind to treatment. A non-blind physician not providing care or ratings will receive real and generate false blood levels to communicate to other investigators for the purpose of titration of the lithium/placebo. Measures for emergency unblinding will be available as well for safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lithium carbonate (Experimental): Lithium carbonate will be initiated at 150 mg per day and increased based on blood levels until a steady blood level between 0.6 and 0.8 meq/L is achieved. Participants will continue at the dose achieved for 2 years with quarterly monitoring.
  Interventions: Drug: Lithium Carbonate
- placebo (Placebo Comparator): Matching placebo will be initiated and increased based on pretend blood levels. Participants will take placebo for 2 years with quarterly monitoring.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Lithium Carbonate — See lithium carbonate arm
  Arms: Lithium carbonate
Drug: Placebo oral capsule — See placebo arm
  Arms: placebo

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia in adults 65 years and older. AD leads to a complete loss of memory and independent function, and presently there is no cure. Many studies suggest that lithium treatment may delay dementia onset or slow its progression. However, more research is needed to understand the extent of its anti-dementia properties if it will be deployed broadly in the general population. This study will examine whether lithium has anti-dementia properties in older adults who have mild cognitive impairment and are at risk of becoming demented.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia in adults 65 years and older. Unchecked, the disease will reach epidemic proportions in the United States and worldwide by 2050, and presently, there is no intervention that has shown a clear effect on AD progression. Over the past several years, there has been increasing interest in re-purposing the use of lithium for diseases involving neurodegeneration. Lithium treatment has been associated with neurogenesis in the hippocampus, up-regulation of important neurotrophic factors such as B-cell lymphoma 2 (Bcl-2) and brain-derived neurotrophic factor (BDNF), and inhibition of glycogen synthase kinase 3 (GSK-3) isoforms α and β. In particular, GSK-3α interacts with gamma-secretase playing a critical role in the conversion of amyloid precursor protein (APP) to amyloid-beta (Aβ); lithium has been shown to reduce Aβ production and memory deficits in AD transgenic mouse models. GSK-3β phosphorylates tau, a critical step in the formation of neurofibrillary tangles, and lithium has been shown to reduce tau phosphorylation in vivo and in vitro. That lithium may alter the AD trajectory is supported by numerous observational reports showing delay of dementia onset in those treated with it. However, the results of the few human lithium trials conducted have been mixed. Additional research is needed to determine whether lithium has a role as an anti-dementia agent. In contrast to previous studies, we will implement an Randomized Controlled Trial (RCT) with a more integrative, comprehensive approach than done before involving state-of-the-art ultra-high field (7T) human Magnetic Resonance Imaging (MRI), neurocognitive assessment, and blood- and Cerebrospinal Fluid (CSF)- based biomarker measurement to investigate the role of lithium as an anti-dementia agent. The specific aim of this pilot-feasibility study is to examine the potential disease modifying properties of lithium in individuals with mild cognitive impairment (MCI) in delaying conversion to dementia. The study will enroll and randomly assign 80 individuals 60 years and older with MCI to take lithium, titrated to a maximally tolerated blood level (0.5 to 0.8 meq/L), or placebo for two years to assess lithium's effects on preserving cognition and delaying conversion to dementia. Participants will receive annual neurocognitive assessment, blood- and CSF-based biomarker measurement, and 7T MRI of structural brain volumes (e.g., hippocampal, total cortical gray). At baseline, all subjects who are able will undergo Positron Emission Tomography (PET) imaging for Aβ. The following hypotheses will be tested: H1: a) Participants randomized to take lithium for two years, compared to placebo, will better maintain cognitive function, primarily in memory, which b) will be associated with changes in biomarkers (e.g., GSK-3β, BDNF). H2: a) Participants randomized to take lithium, compared to placebo, will have larger hippocampal volumes and lower total gray matter thinning, which b) will be associated with changes in biomarkers and c) better cognitive function, primarily in memory. The exploratory aim examines whether lithium is related to additional markers of enhanced brain integrity (e.g., lower level of microbleeds, higher white matter integrity, better network connectivity, or decreased CSF phospho tau levels).

The following amendments were made with entering the results to correct mistakes in the original registration:

1. Primary Outcome 6 was corrected to Cerebral Cortical Gray Matter Volume.
2. Primary Outcome 7 was correct to Hippocampal Volume.
3. The outcome measure "Change From Baseline Brain Integrity Measures Over 2 Years as Measured by Structural Imaging (7T MRI)" was corrected to Other Pre-Specified Outcome Measure(s).
4. The outcome measure "NIH Toolbox" was corrected to PostHoc Outcome Measure(s).

ELIGIBILITY:
Inclusion Criteria:

1. 60 years or older
2. Diagnosis of Mild Cognitive Impairment

Exclusion Criteria:

1. Major psychiatric illness (mild psychiatric illness may be included)
2. Major neurologic illness (e.g., multiple sclerosis)
3. Contraindication to lithium (e.g., renal insufficiency)
4. Unable to complete neuropsychological testing due to non-remediable impairment (e.g., blindness)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Gildengers, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared with the National Cell Repository for Alzheimer's Disease (NCRAD).

REFERENCES:
- [Derived] Gildengers AG, Ibrahim TS, Zeng X, Aizenstein HJ, Alkhateeb SK, Anderson SJ, Chu C, Diaz JL, Emanuel JE, Karikari TK, Li J, Lopez OL, Lopresti BJ, Royse SK, Sajewski AN, Santini T, Weinstein AM, Wu M, Butters MA. The LATTICE Study: Design of a pilot feasibility randomized controlled trial of lithium to delay cognitive decline in mild cognitive impairment. Alzheimers Dement (N Y). 2025 Jun 11;11(2):e70112. doi: 10.1002/trc2.70112. eCollection 2025 Apr-Jun. PMID 40501510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following Data and Safety Monitoring Board approval 9/1/2017, the first participant enrolled 2/2/2018, and last enrolled 8/29/2022. Recruitment involved senior centers, education classes, communities, housing, internet methods, University of Pittsburgh Alzheimer's Disease Research Center partnerships, primary care practices, former participants. During the pandemic, internet/print ads replaced in-person activities.
Groups:
- Lithium Carbonate: Lithium carbonate will be initiated at 150 mg per day and increased based on blood levels to a steady blood level between 0.6 and 0.8 meq/L or the maximum tolerated dose based on side effects if lower. Participants will continue at the dose achieved for 2 years with quarterly monitoring.
  Lithium Carbonate: See lithium carbonate arm
Period: Overall Study
Arm/Group | Lithium Carbonate | Placebo
Started | 41 | 42
Completed | 41 | 39
Not Completed | 0 | 3
Not completed — Did not start study medication | 0 | 3

BASELINE CHARACTERISTICS:
Population: Three participants in the placebo arm withdrew consent after randomization, but prior to initiating the study medication and are excluded from the baseline sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Carbonate | Placebo | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Pooled mean and pooled standard deviation.
  years | 72.93 (8.77) | 71.22 (6.47) | 72.10 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 41 | 38 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 38 | 33 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education (years) [Mean (Standard Deviation); unit: years] | 15.46 (2.66) | 16.54 (1.8) | 15.99 (2.33)
Amyloid-beta [Count of Participants; unit: Participants] — Positron Emission Tomography (PET)-amyloid imaging classification amyloid-beta positive or negative. PET-amyloid imaging is a specialized brain scan that can detect abnormal protein deposits called amyloid-beta plaques, which are a hallmark of Alzheimer's disease. Amyloid-positive: Significant amyloid plaques are present in the brain. Amyloid-negative: Little to no amyloid plaques are detected.
  Participants
    Amyloid-beta negative | 27 | 27 | 54
    Amyloid-beta positive | 11 | 10 | 21
    Amyloid-beta unknown | 3 | 2 | 5
Mild Cognitive Impairment [Count of Participants; unit: Participants] — Mild Cognitive Impairment (MCI) means having memory or thinking problems that are more than normal aging but not severe enough to be dementia. Amnestic MCI - primarily affects memory. Non-amnestic MCI - affects thinking skills other than memory.
  Participants
    Amnestic | 34 | 28 | 62
    Not Amnestic | 7 | 11 | 18
APOE e4 allele [Count of Participants; unit: Participants] — The Apolipoprotein E (APOE) e4 allele is a specific version of the APOE gene that significantly increases your risk of developing Alzheimer's disease. Carrier means that the participant has at least one copy of the gene.
  Participants
    Non-carrier | 26 | 26 | 52
    Carrier | 15 | 13 | 28
Framingham Stroke Risk Profile [Mean (Standard Deviation); unit: percentage] — The Framingham Stroke Risk Profile (FSRP) estimates 10-year stroke probability using age, sex, blood pressure, diabetes, smoking, cardiovascular disease, and atrial fibrillation. Scores range from 0.50% to 95.71%. Higher scores indicate greater stroke risk, helping guide prevention strategies and treatment decisions.
  percentage | 13 (12) | 11 (12) | 12 (12)
Cumulative Illness Rating Scale-Geriatric [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale-Geriatric (CIRS-G) measures medical illness burden across 14 organ systems, each scored 0-4 (none to extremely severe). Total scores range from 0 to 56. Higher scores indicate greater comorbidity burden and illness severity, predicting mortality and healthcare outcomes in older adults.
  units on a scale | 11.07 (4.67) | 9.9 (3.61) | 10.50 (4.2)
Creatinine [Mean (Standard Deviation); unit: mg/dL] — Serum creatinine is a blood test measuring creatinine. Normal levels are roughly 0.6-1.2 mg/dL for adults. Higher levels indicate decreased kidney function or kidney disease. It is used to assess kidney health and calculate estimated glomerular filtration rate (eGFR).
  mg/dL | 0.84 (0.16) | 0.92 (0.14) | 0.88 (0.15)
Glomerular Filtration Rate (GFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Glomerular filtration rate (GFR) measures how well kidneys filter blood, indicating kidney function. Normal GFR is 90+ mL/min/1.73m². Values 60-89 suggest mild decrease, 30-59 moderate decrease, 15-29 severe decrease, and <15 kidney failure. Estimated GFR (eGFR) is calculated from serum creatinine.
  mL/min/1.73m^2 | 84.23 (11.74) | 77.95 (13.11) | 81.17 (12.74)
Medication count [Mean (Standard Deviation); unit: Number of medications] — Total number of medications prescribed to the participant.
  Number of medications | 7.78 (5.22) | 6.64 (4.84) | 7.23 (5.04)
Anticholinergic Burden [Mean (Standard Deviation); unit: units on a scale] — Anticholinergic burden measures cumulative effects of medications blocking acetylcholine. The scale ranges from 0 (no burden) to 5+ (high burden), with each medication contributing 0-3 points based on anticholinergic activity. Scores ≥3 are clinically significant, warranting medication review due to increased risk of cognitive impairment, falls, and other anticholinergic side effects. Total score is the sum of individual medication scores (0-3 each). No maximum total score exists.
  units on a scale | 2.53 (2.39) | 2.34 (2.85) | 2.44 (2.61)
Physical Activity Scale for the Elderly (PASE) [Mean (Standard Deviation); unit: units on a scale] — The Physical Activity Scale for the Elderly (PASE) measures self-reported physical activity in adults 65+ across leisure, household, and occupational activities over 7 days. Scores range from 0 to 793 with typical scores ranging 0 to 400+. Higher scores indicate greater physical activity levels and better health outcomes.
  units on a scale | 117.01 (73.65) | 90.20 (50.91) | 103.77 (64.47)
Patient Health Questionnaire-9 item (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a 9-item depression screening tool. Scores range from 0-27, with each item rated 0-3. Higher scores indicate more severe depression: 0-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depression.
  units on a scale | 3.88 (3.27) | 3.49 (3.46) | 3.69 (3.35)
Brief Visual Memory Test Revised (BVMT-R) [Mean (Standard Deviation); unit: units on a scale] — The Brief Visuospatial Memory Test-Revised (BVMT-R) assesses visual memory using 6 geometric figures learned over 3 trials, then delayed recall after 25 minutes. Each trial has a maximum of 12 points, with Total Recall scores ranging 0-36 and Delayed Recall 0-12. Higher scores indicate better visual memory and learning ability. Delayed Recall score is presented. Population: One participant in Group lithium did not receive the BVMT-R and CVLT-II because she had substantial familiarity with those tests.
  units on a scale
    number analyzed (Participants) | 40 | 39 | 79
    (all) | 6.23 (3.11) | 6.56 (2.86) | 6.39 (2.98)
California Verbal Learning Test 2nd edition (CVLT-II) [Mean (Standard Deviation); unit: units on a scale] — The California Verbal Learning Test 2nd Edition (CVLT-II) assesses verbal learning and memory using a 16-word list learned over 5 trials, plus delayed recall and recognition. Total Learning scores range 0-80 (16 words × 5 trials), delayed recall 0-16. Higher scores indicate better verbal learning and memory performance. Delayed recall score is presented. Population: One participant in Group lithium did not receive the BVMT-R and CVLT-II because she had substantial familiarity with those tests.
  units on a scale
    number analyzed (Participants) | 40 | 39 | 79
    (all) | 7.95 (3.4) | 7.90 (3.9) | 7.92 (3.63)
Preclinical Alzheimer's Cognitive Composite (PACC) [Mean (Standard Deviation); unit: Z-score] — The Preclinical Alzheimer's Cognitive Composite (PACC) combines tests assessing episodic memory, executive function, and global cognition to detect early cognitive decline before clinical symptoms appear. Higher scores indicate better cognitive performance. A Z-score of 0 represents the population mean, while Z-scores of ±1 capture approximately 68% of the data around the mean and Z-scores of ±2 capture approximately 95% of the data in a normal distribution. Population: Three Group placebo participants had missing data, preventing calculation of their PACC scores.
  Z-score
    number analyzed (Participants) | 41 | 36 | 77
    (all) | -0.36 (3.59) | 0.41 (3.16) | 0.00 (3.39)
Hippocampal volume [Mean (Standard Deviation); unit: mm^3] — Hippocampal volume measures the size of the hippocampus, a brain region crucial for memory formation and learning. Smaller volumes indicate atrophy and are associated with memory impairment, Alzheimer's disease, depression, and aging. These values are not corrected for age, sex, and intracranial volume. Population: 18 participants were unable to complete neuroimaging or images were not analyzable.
  mm^3
    number analyzed (Participants) | 33 | 29 | 62
    (all) | 7387 (1293) | 7199 (801) | 7299 (1087)
Cerebral Cortical Gray Matter [Mean (Standard Deviation); unit: mm^3] — Cerebral cortical gray matter volume measures the total amount of gray matter (neuron cell bodies, dendrites, synapses) in the brain's outer cortex. Reduced volumes are associated with aging, neurodegeneration, and cognitive decline. These values are not corrected for age, sex, and intracranial volume. Population: 18 participants were unable to complete neuroimaging or images were not analyzable.
  mm^3
    number analyzed (Participants) | 33 | 29 | 62
    (all) | 416997 (51634) | 410702 (40439) | 414053 (46468)
Brain derived neurotrophic factor [Mean (Standard Deviation); unit: Log transformed number of molecules] — Brain-Derived Neurotrophic Factor (BDNF) supports neuron survival and growth; reduced levels linked to neurodegeneration. Nucleic Acid-Linked Immuno-Sorbent Assay (NULISA) measures BDNF using nucleic acid-tagged antibody pairs recognizing different BDNF epitopes. Sequential capture/purification via polyA/biotin tails, then ligation and next-generation sequencing quantification achieves attomolar sensitivity alongside hundreds of other proteins. Population: Seven participants had missing BDNF values at baseline due to insufficient blood samples or for failing quality control.
  Log transformed number of molecules
    number analyzed (Participants) | 36 | 37 | 73
    (all) | 14.61 (0.83) | 14.41 (1.47) | 14.51 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test II
Description: California Verbal Learning Test II. Long-delay free recall. Scores range from 0 - 16; higher means better.
Time Frame: Year 1 and Year 2
Population: Intention-to-treat analysis; all randomized participants were included regardless of study completion or protocol adherence.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 40 | 39
units on a scale
  Year 1: number analyzed (Participants) | 37 | 31
  Year 1 | 6.9 (4.0) | 6.2 (4.6)
  Year 2: number analyzed (Participants) | 37 | 31
  Year 2 | 6.46 (3.97) | 5.10 (4.54)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.048, Mixed Models Analysis; treatment x time interaction coefficient = 0.69

2. Primary Outcome: Brief Visuospatial Memory Test - Revised
Description: Brief Visuospatial Memory Test - Revised. Delayed Recall. Scores range from 0 - 12; higher means better.
Time Frame: Year 1 and Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 40 | 39
units on a scale
  Year 1: number analyzed (Participants) | 38 | 31
  Year 1 | 5.97 (3.2) | 5.9 (3.1)
  Year 2: number analyzed (Participants) | 36 | 31
  Year 2 | 5.69 (3.4) | 6.19 (3.73)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.78, Mixed Models Analysis; treatment x time interaction coefficient = -0.08835

3. Primary Outcome: Preclinical Alzheimer Cognitive Composite Composed of Memory and Other Cognitive Tests
Description: Cognitive testing measures with a composite of memory, executive function, processing speed, activities of daily living, and general cognition tests. Values are Z-scores. Higher values mean better cognition. A Z-score of 0 represents the population mean, while Z-scores of ±1 capture approximately 68% of the data around the mean and Z-scores of ±2 capture approximately 95% of the data in a normal distribution.
Time Frame: Year 1 and Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 41 | 36
Z-score
  Year 1: number analyzed (Participants) | 35 | 25
  Year 1 | 0.10 (4.3) | 0.43 (3.7)
  Year 2: number analyzed (Participants) | 37 | 28
  Year 2 | -0.67 (5.67) | -0.19 (4.04)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.80, Mixed Models Analysis; treatment x time interaction coefficient = 0.08738

4. Primary Outcome: Glycogen Synthase Kinase-3 Beta (GSK-3β) Activity
Description: Values of blood-based biomarkers
Time Frame: Year 1 and Year 2
Population: The researchers could not evaluate GSK-3β as commercial assays failed to reliably measure its activity in plasma.
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Brain-derived Neurotrophic Factor
Description: Brain-Derived Neurotrophic Factor (BDNF) supports neuron survival and growth; reduced levels linked to neurodegeneration. Nucleic Acid-Linked Immuno-Sorbent Assay (NULISA) measures BDNF using nucleic acid-tagged antibody pairs recognizing different BDNF epitopes. Sequential capture/purification via polyA/biotin tails, then ligation and next-generation sequencing quantification achieves attomolar sensitivity alongside hundreds of other proteins.
Time Frame: Year 1 and Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log transformed number of molecules
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 41 | 39
Log transformed number of molecules
  Year 1: number analyzed (Participants) | 37 | 26
  Year 1 | 14.5 (1.02) | 14.1 (1.71)
  Year 2: number analyzed (Participants) | 38 | 31
  Year 2 | 14.5 (0.90) | 14.3 (1.33)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.93, Mixed Models Analysis; treatment x time interaction coefficient = 0.012

6. Primary Outcome: Cerebral Cortical Gray Matter Volume
Description: Cerebral cortical gray matter volume as measured by structural imaging (7T MRI) corrected for age, sex, and intracranial volume
Time Frame: Year 1 and Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 33 | 29
mm^3
  Year 1: number analyzed (Participants) | 31 | 23
  Year 1 | 412951 (24063) | 405236 (16950)
  Year 2: number analyzed (Participants) | 28 | 22
  Year 2 | 411270 (27271) | 402212 (19033)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.78, Mixed Models Analysis; treatment x time interaction coefficient = -351.8

7. Primary Outcome: Hippocampal Volume
Description: Hippocampal volume values as measured by structural imaging (7T MRI) corrected for age, sex, and intracranial volume
Time Frame: Year 1 and Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 33 | 29
mm^3
  Year 1: number analyzed (Participants) | 31 | 23
  Year 1 | 7352 (847) | 7118 (816)
  Year 2: number analyzed (Participants) | 28 | 22
  Year 2 | 7369 (812) | 6884 (922)
Statistical Analysis 1: Comparison: Lithium Carbonate vs Placebo; Test type: Superiority; p = 0.087, Mixed Models Analysis; treatment x time interaction coefficient = 58.95

8. Secondary Outcome: Cerebrospinal Fluid Phospho Tau Level (CSF)
Description: Cerebrospinal fluid phospho tau levels
Time Frame: Year 1 and Year 2
Population: CSF collection was not performed due to insufficient participant consent for lumbar puncture procedures.
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Brain Integrity as Measured by Structural Imaging (7T MRI)
Description: Exploratory analyses of additional measures of brain integrity, such as lower level of microbleeds, higher white matter integrity, or better network connectivity
Time Frame: Year 1 and Year 2
Reporting Status: Not Posted

10. Post Hoc Outcome: NIH Toolbox
Description: NIH Toolbox performance
Time Frame: Year 1 and Year 2
Population: Valid NIH Toolbox cognitive composite scores were available for only one participant at baseline and 2-year follow-up due to two factors: 1) Coronavirus Disease 2019 (COVID-19) protocol changes required remote administration, for which composite scores are not provided due to unknown validity effects, and 2) composite scores are not available for participants aged 86+. The pandemic timing caused additional missing data, leaving only one participant with complete data across timepoints.
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: At weekly titration visits until participants achieved a steady dose within target range or the maximum tolerated dose, then at monthly/quarterly/annual visits thereafter during their 2 year treatment period. Additional data was collected if participants contacted study staff outside of these visits and reported adverse events, if an extra visit was necessary for added clinical monitoring, or if study staff identified serious adverse events when reviewing medical records.
Arm/Group | Lithium Carbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 1/39
Serious Adverse Events (participants affected / at risk) | 12/41 | 9/39
Other Adverse Events (participants affected / at risk) | 41/41 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=41) | Placebo (N=39)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Hemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Vasovagal Episode (Vascular disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Rheumatoid lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — Includes flare up and respiratory failure
Nausea and left arm pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dislocation of right hip (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Recurrence of atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Shortness of breath (Cardiac disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (2) | 0 (0) — Include acute kidney injury and weakness
Fever and shortness of breath (Infections and infestations) | 1 (1) | 0 (0)
Leg pain and swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg wounds (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Etadolac related ischemic colitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infectious aortitis (Infections and infestations) | 1 (1) | 0 (0)
Bleeding stomach ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) — Includes recurrence
Neck surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Fall, fracture of right hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shortness of breath, pedal edema, pulmonary embolism, acute atrial flutter with RVR on chronic CHF (Cardiac disorders) | 1 (1) | 0 (0) — Shortness of breath, pedal edema, pulmonary embolism, acute atrial flutter with rapid ventricular response on chronic congestive heart failure.
Frequent falls (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bilateral hip and leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Confusion and shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radiation treatment of malignant skin neoplasm and osteomyelitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Total knee athroscopy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Left or right
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=41) | Placebo (N=39)
Increased creatinine (Renal and urinary disorders) | 12 (16) | 12 (21)
Tremor (Nervous system disorders) | 10 (13) | 6 (18)
Sleepiness (General disorders) | 10 (19) | 9 (12)
Tiredness (General disorders) | 12 (19) | 6 (9)
Increased urinary frequency (Renal and urinary disorders) | 4 (9) | 6 (14)
Diarrhea (Gastrointestinal disorders) | 12 (21) | 6 (11)
Dizziness (General disorders) | 5 (10) | 6 (9)
Dry mouth (General disorders) | 4 (7) | 3 (6)
Weight gain (Metabolism and nutrition disorders) | 7 (9) | 4 (5)
Increase TSH value (Endocrine disorders) | 7 (7) | 3 (5)
Unsteadiness (General disorders) | 5 (8) | 3 (7)
Edema (Vascular disorders) | 5 (11) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 2 (4) | 4 (6)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (3)
Increased calcium value (Blood and lymphatic system disorders) | 5 (7) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (4)
Indigestion (Gastrointestinal disorders) | 1 (2) | 2 (3)
Pedal edema (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
Concentration difficulties (General disorders) | 3 (3) | 2 (2)
Memory difficulties (Nervous system disorders) | 2 (2) | 1 (1)
Increased thirst (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (3) | 1 (1)
Headache (General disorders) | 5 (11) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Mouth ulcers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Metallic taste (General disorders) | 1 (1) | 0 (0)
Electrolyte abnormality (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypnogogic hallucination (Nervous system disorders) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 4 (5) | 1 (1)
Falls, recurrent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accommodation Disturbance (Eye disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (2) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (8) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (General disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Facial nerve palsy (Nervous system disorders) | 1 (2) | 0 (0)
Facial pain (General disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heaviness in limbs (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hives (General disorders) | 0 (0) | 1 (2)
Hot flashes (General disorders) | 1 (2) | 0 (0)
Hungriness (General disorders) | 0 (0) | 1 (1)
Increased dream activity (Psychiatric disorders) | 1 (1) | 2 (3)
Increased sleep duration (Psychiatric disorders) | 1 (1) | 0 (0)
Inner unrest (General disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 2 (2) | 6 (10)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1)
Itchiness (General disorders) | 1 (2) | 1 (2)
Leg cramps (General disorders) | 0 (0) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Mechanical fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Micturation difficulty (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Night sweats (General disorders) | 1 (1) | 1 (1)
Palpitations (General disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reduced emotional flattening (Psychiatric disorders) | 0 (0) | 1 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Somniloquy (General disorders) | 0 (0) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stuttering (Psychiatric disorders) | 1 (2) | 0 (0)
Twitching in sleep (Psychiatric disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The results presented are preliminary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03185208/Prot_SAP_000.pdf